CLINICAL TRIAL: NCT05736146
Title: Validating Blood Biomarkers of Brain Immune and Metabolic Dysfunction in Gulf War Illness
Brief Title: Validating Gulf War Illness Blood Biomarkers
Status: Recruiting | Type: Observational
Sponsor: Roskamp Institute Inc. (Other)
Collaborators: Boston University (Other); Palo Alto Veterans Institute for Research (Other); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: RI-GWI-003
Record Dates: First submitted 2023-02-09; First posted 2023-02-21 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2024-11

CONDITIONS: Gulf War Syndrome; Gulf War Illness
Keywords: Gulf War; APOE
MeSH Terms: conditions — Persian Gulf Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be analyzed for lipids, proteins, DNA, RNA and breakdown products to identify biomarkers for GWI.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Case: GWI: This group includes participants who served in the Gulf War during 1990 -1991 and have Gulf War Illness based on either the Kansas or CDC symptom criteria.
- Control: This group includes participants who served in the Gulf War during 1990 -1991 and have no symptoms of Gulf War Illness based on both the Kansas and CDC symptom criteria.

SUMMARY:
The investigators goals are to identify blood lipids/metabolites that correlate with cognitive decline in the presence of the APOE ε4 allele among veterans with GWI. To determine the effect of dietary, medical and biological factors that influence lipid and metabolites in blood from GW veterans. To identify blood lipid/metabolite profiles that correlate with bioenergetics deficits and glial activation in the brains of GWI. To validate blood biomarker signatures of GWI using APOE genotyping and blood lipids/metabolites that correlate with the CNS dysfunction in GWI.

DETAILED DESCRIPTION:
Nearly 30 years later, veterans with Gulf War Illness (GWI) continue to suffer from this persistent and debilitating illness, which remains difficult to diagnose due to the heterogeneity of clinical presentation and the complexity of biological responses to hazardous chemicals to which GW veterans were exposed during the 1990-1991 Gulf War (GW). Brain imaging studies of veterans with GWI and pre-clinical animal studies of rodents with GWI show that impaired bioenergetics and inflammation can be attributed to the atrophy of the axonal white matter tracts that link the cortical gray matter regions, and the alterations of lipid/metabolite levels. The investigators recent work shows that disturbed lipid profiles in the brain and blood after GW pesticide exposure in rodents accompany neurobehavioral and bioenergetics deficits and inflammation. The mechanisms of neurotoxicity after pesticide exposure include increases in the inactivation of lipid metabolizing enzymes. This may consequently result in accumulation of lipids in the body compartments that limit their availability for use as energy substrates, contributing to bioenergetic impairments and inflammation. These metabolic changes have also been linked to individuals who possess the apolipoprotein E (APOE) ε4 allele, a risk factor of aging related cognitive decline and neurodegenerative conditions, such as Alzheimer's disease (AD). Several studies have shown a correlation between lipid transport deficits and presence of the ε4 allele. The identification of specific lipids/metabolites and the APOE ε4 allele as important biomarkers of GWI would serve to objectively assess the brain pathology of GWI and identify subgroups of GWI based on symptom patterns and GW exposures.

ELIGIBILITY:
Inclusion Criteria:

1. Age 35 years or older.
2. For GWI cases, served in the 1990-1991 Gulf War as active duty, national guard, or reserves and meet criteria for the CDC Chronic Multisymptom Illness (CMI) GWI definition or Kansas GWI definition.
3. For controls, must be a veteran in the same age range as those veterans with GWI as defined above.
4. Ability to understand written and spoken English or availability of a legal representative who can understand written or spoken English. Participants and caregiver/informants must be able to read, write and speak the language in which psychometric tests are provided with visual and auditory acuity (corrected) sufficient to allow for accurate testing.

Exclusion Criteria:

1. Diagnosed or being treated by a physician for any of the following (Steele et al, 2000) and deemed clinically significant per the discretion of the PI:

   1. Cancer (except for non-melanoma skin cancers)
   2. Chronic infectious disease
   3. Problems resulting from postwar injuries.
   4. Liver disease
   5. Lupus
   6. Multiple sclerosis
   7. Stroke
   8. Serious psychiatric condition (those associated with psychosis and/or for which the respondent had been hospitalized since 1991).
   9. Dementia or any type of Parkinson's disease (PD).
2. Hospitalized in the last 5 years for alcohol or drug dependence, depression, or post-traumatic stress disorder (PTSD).
3. Female subject is either pregnant or nursing.

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Veterans who served in the Gulf War during 1990 to 1991.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-06-30 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Validate Blood Biomarkers | 2022-2024
  To validate blood biomarker signatures of GWI using APOE genotyping and blood lipids/metabolites that correlate with the CNS dysfunction in GWI.
Identify Blood/Lipid Profiles | 2022-2024
  To identify blood lipid/metabolite profiles that correlate with bioenergetics deficits and glial activation in the brains of GWI.
Effect of Dietary, Medical and Biological Factors | 2022-2024
  To determine the effect of dietary, medical and biological factors that influence lipid and metabolites in blood from GW veterans.
Metabolites Correlating with Cognitive Decline | 2022-2024
  To identify blood lipids/metabolites that correlate with cognitive decline in the presence of the APOE ε4 allele among veterans with GWI.

CONTACTS AND LOCATIONS:
Overall Officials: Laila Abdullah, Ph.D., Principal Investigator — The Roskamp Institute; Michael Hoffmann, MD, Principal Investigator — The Roskamp Institute; Kim Sullivan, Ph.D, Principal Investigator — Boston University; Maheen Adamson, Ph.D., Principal Investigator — Palo Alto Veterans Institute of Research
Locations (3):
- United States (3):
  - Palto Alto Veterans Institute for Research, Palo Alto, California
  - The Roskamp Institute, Sarasota, Florida
  - Boston University, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Roskamp Institute Home Page — http://www.roskampinstitute.org/